CLINICAL TRIAL: NCT06946667
Title: Pathogen Resistance Characteristics and Development of a Combined Diagnostic Model Using Hs-CRP, HBP, NGAL, and ADPN for Postoperative Urinary Tract Infections in Patients With Kidney Stones
Brief Title: Resistance Characteristics and Development of Diagnostic Model for Postoperative UTI in Patients With Kidney Stones
Status: Completed | Type: Observational
Sponsor: Xingxin Jiang (Other Government)
Responsible Party: Sponsor-Investigator, Xingxin Jiang, Principal Investigator, Suzhou Hospital of Integrated Traditional Chinese and Western Medicine
Organization: Suzhou Hospital of Integrated Traditional Chinese and Western Medicine (Other Government)
Other Study IDs: No. 2025-008
Record Dates: First submitted 2025-04-06; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-01

CONDITIONS: Urinary Tract Infection Complicated; Kidney Stones; Antimicrobial Resistance
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the UTI group: Midstream clean-catch urine samples from patients in the UTI group were collected for pathogen identification and antimicrobial susceptibility testing.
  Interventions: Other: the UTI group
- the Non-UTI group: Midstream clean-catch urine samples from patients in the UTI group were collected for pathogen identification and antimicrobial susceptibility testing.
  Interventions: Other: the Non-UTI group

INTERVENTIONS:
Other: the UTI group — Laboratory parameters, including WBC, NLR, NEU, hs-CRP, HBP, NGAL, and ADPN levels, were measured. Midstream clean-catch urine samples from patients in the UTI group were collected for pathogen identification and antimicrobial susceptibility testing.
  Groups: the UTI group
Other: the Non-UTI group — Laboratory parameters, including WBC, NLR, NEU, hs-CRP, HBP, NGAL, and ADPN levels, were measured. Midstream clean-catch urine samples from patients in the UTI group were collected for pathogen identification and antimicrobial susceptibility testing.
  Groups: the Non-UTI group

SUMMARY:
The combined detection of HBP, ADPN, NGAL, and hs-CRP enables the construction of a highly efficient diagnostic model, offering a novel strategy for early infection identification and risk stratification after surgery.

DETAILED DESCRIPTION:
This study investigated pathogen distribution, antimicrobial resistance, and the diagnostic utility of biomarkers (hs-CRP, HBP, NGAL, ADPN) for Urinary Tract Infections (UTI) after kidney stone surgery. A total of 130 patients with kidney stones, treated between February 2021 and December 2024, were included in this study. Based on the occurrence of postoperative UTIs, they were categorized into the UTI group (n=41) and the Non-UTI group (n=89). Laboratory parameters, including WBC, NLR, NEU, hs-CRP, HBP, NGAL, and ADPN levels, were measured. Midstream clean-catch urine samples from patients in the UTI group were collected for pathogen identification and antimicrobial susceptibility testing. Pearson correlation analysis was performed to assess the relationships among these biomarkers, ROC curve analysis was conducted to evaluate diagnostic performance, and logistic regression analysis was used to identify independent risk factors for postoperative infections.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Diagnosis of urinary calculi confirmed by CT, X-ray, or ultrasound;
3. Complete clinical data available. -

Exclusion Criteria:

1. Presence of active UTI or other infections prior to surgery;
2. Coexisting urological disorders (e.g., bladder cancer, neurogenic bladder);
3. Prolonged use of immunosuppressants or antibiotics (>2 weeks). -

Ages: 44 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: A total of 130 patients diagnosed with kidney stones and treated at our hospital between February 2021 and December 2024 were enrolled in this study. Based on the presence of postoperative UTI, patients were categorized into the UTI group (n=41) and the Non-UTI group (n=89). The mean age of patients in the UTI group was 52.76±8.49 years, comprising 24 males and 17 females, whereas the Non-UTI group had a mean age of 53.03±7.12 years, including 43 males and 46 females.
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Pathogen Resistance Characteristics and Development of a Combined Diagnostic Model Using hs-CRP, HBP, NGAL, and ADPN for Postoperative Urinary Tract Infections in Patients with Kidney Stones | 10 weeks
  Postoperative UTI in kidney stone patients are primarily caused by Gram-negative bacteria with high resistance. Combined detection of hs-CRP, HBP, NGAL, and ADPN significantly improves diagnostic accuracy. HBP, NGAL, and ADPN serve as early predictive markers for postoperative infection, providing a reference for clinical practice.

CONTACTS AND LOCATIONS:
Locations (1):
- Suzhou Hospital of Integrated Traditional Chinese and Western Medicine, Suzhou, Jiangsu, China